CLINICAL TRIAL: NCT03572270
Title: Evaluation of the Potential Impact of HIV and Its Treatments on Ovarian Reserve: Prospective Study
Brief Title: HIV and Ovarian Reserve
Acronym: VIHRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-391; 2017-A03469-44 (Other: 2017-A03469-44)
Record Dates: First submitted 2018-05-29; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: HIV; Infertility
Keywords: HIV; Ovarian reserve; Fertility preservation; Anti HIV agents
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Masking Description: No masking
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- case (Experimental): PLWH
  Interventions: Diagnostic Test: AMH test; Diagnostic Test: pelvic ultrasound
- control (Other): HIV negative women, going to medically assisted procreation consultation for male infertility
  Interventions: Diagnostic Test: AMH test; Diagnostic Test: pelvic ultrasound

INTERVENTIONS:
Diagnostic Test: AMH test — Blood test and pelvic ultrasound are performed at each visit to evaluate ovarian reserve
Diagnostic Test: pelvic ultrasound — Blood test and pelvic ultrasound are performed at each visit to evaluate ovarian reserve

SUMMARY:
Recent evidence suggests a decline in fertility of persons living with HIV (PLWH) (delayed pregnancies, sponteanous abortions, especially when patients receive an antiretroviral therapy, early menopause, amenorrhea and anovulatory cycles) with a possible decrease in ovarian reserve. However, indications of fertility preservation by freezing oocytes are nevertheless not clearly identified.

The objective of this study is to evaluate the ovarian reserve before and after the implementation of antiretroviral treatment in PLWH for whom the diagnosis of HIV has just been made.

DETAILED DESCRIPTION:
This is a monocentric prospective cohort study with minimal risk and constraints. Ovarian reserve is compared between two groups: 30 PLWH, at time of diagnosis and 6, 12 and 18 months after initiation of an antiretroviral therapy, and 30 HIV negative women attending medically assisted procreation consultation for male infertility, age, BMI and smoking habits matched.

ELIGIBILITY:
Inclusion Criteria:

* For every participant :
* woman aged 18 to 37
* covered by social security
* able to give an informed consent

Case group only :

* diagnosis of HIV infection during the 3 months before inclusion
* concomitant initiation of an antiretroviral therapy with integrase inhibitors and nucleoside analogues

Control group only :

* assisting medically assisted procreation consultation for male infertility
* matching case subjects with age, BMI and smoking habits

Exclusion Criteria:

* For every participant :
* current pregnancy
* condition or associated treatment that may have an impact on fertility
* premature ovarian failure
* polycystic ovary syndrome
* endometriosis

Control group only :

- suspected HIV infection

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
change from inclusion visit AMH level at 18 months | M0 (inclusion visit) and M18 (after 18 months)
  blood test to evaluate ovarian reserve thanks to AMH

SECONDARY OUTCOMES:
antral follicle count | Month 0 (inclusion visit), Month 6 (after 6 months), Month12 (after one year), Month18 (after 18 months)
  pelvic ultrasound to evaluate ovarian reserve thanks to antral follicle count
estradiol, lutenizing hormone and follicle-stimulating hormone test | Month 0 (inclusion visit), Month 6 (after 6 months), Month 12 (after one year), Month18 (after 18 months)
  blood test

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRUGNON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France